CLINICAL TRIAL: NCT03428425
Title: A Study of HIPEC Plus Apatinib and S-1 Conversion Therapy for Gastric Cancer With Positive Exfoliative Cancer Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRA-G02
Record Dates: First submitted 2018-02-01; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib paclitaxel S-1 (Experimental)
  Interventions: Drug: paclitaxel apatinib S-1

INTERVENTIONS:
Drug: paclitaxel apatinib S-1 — HIPEC: 43℃, 60min. the drug is paclitaxel : 70mg/m2 d1 d3 d5, The interval is not less than 24h , A total of three times.
  apatinib：500mg qd po, 28 days is a cycle.preoperative 2 cycles, 2 cycles after surgery.
  S-1： According to the body surface area, BSA <1.25m2，40mg bid; 1.25m2≤BSA≤1.5m2，50mg bid; BSA >1.5m2, 60mg bid. Take the medicine twice daily for 2 weeks, then suspend for 1 week. preoperative 3 cycles, 3 cycles after surgery

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of HIPEC plus apatinib and S-1 in the conversion therapy of gastric cancer with positive exfoliative cancer cells

ELIGIBILITY:
Inclusion Criteria:

* 1. Untreated (e.g. chemotherapy, radiotherapy and other antitumor therapy); 2. Age:18 to 70 years old; 3. Man or female (except pregnant and lactating women); 4. Conﬁrmed to gastric adenocarcinoma; 5. Proven gastric cancer of T stage was T3 and T4, and no distant metastasis was observed. The exfoliative cancer cells detection in peritoneal washes was positive; 6. Blood cell count has to meet the following certeria: WBC≥3.5×109/L; ANC≥1.5×109/L; PLT≥100×109/L; HB≥90g/L; 7. Liver/kidney function has to meet the following certeria: ALT and AST≤2.5×ULN TBIL<1.5×ULN； Serum creatinine ≤1.5×ULN; 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; 9. Participants were willing to join in this study, good adherence and written informed consent.

Exclusion Criteria:

- 1. Patients with other malignant tumors within 5 years; 2. Metastasis was found to be visible to the naked eye; 3. It has serious or uncontrolled heart diseases and infections (Including atrial fibrillation, angina pectoris, cardiac insufficiency, ejection fraction less than 50%, poor-controlled hypertension and so on); 4. History of psychiatric drugs abuse and can't quit or patients with mental disorders; 5. Patients with severe or uncontrollable mental illness; 6. Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (+ +).Has melena and hematemesis in two months; 7. Pregnant or lactating women; 8. It have serious harm to the patient's safety or affect the patients who have completed the research.

9. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
R0-resection rate | within 3 weeks after surgery
  There was no residual by the microscope
Conversion to negative rate | within 3 weeks after surgery
  Exfoliative cytology positive gastric cancer conversion to negative rate

SECONDARY OUTCOMES:
Overall survival (OS) | 5years
  Baseline to measured date of death from any cause
Progression free survival (PFS) | 5years
  Baseline to measured date of progression or death from any cause
Adverse events | 5 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.The number of Participants with adverse events will be recorded at each treatment visit